CLINICAL TRIAL: NCT01570335
Title: The SBAR Effect on Safety Attitudes in the Perinatal Department
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 101010-E
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2013-03

CONDITIONS: Fetal Distress
Keywords: SBAR,; SAQ,; Team Resource Management
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The aim of this study is to analyze the impact of SBAR by the SAQ questionnaire in the perinatal department.

ELIGIBILITY:
Inclusion Criteria:

* All Physicians and Nurses in the Perinatal Department

Exclusion Criteria:

* nil

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Physicians and Nurses in the Perinatal Department
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes of patient safety attitude after introducing SBAR | 6 month
  Changes of patient safety attitude after introducing SBAR in the perinatal ward

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan